CLINICAL TRIAL: NCT00217971
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Dronabinol in the Treatment of Marijuana Addiction
Brief Title: Dronabinol Treatment for Marijuana Addiction
Acronym: MARINOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4886-NIDA-09236-11; P50DA009236 (NIH); P50DA009236-11 (NIH); DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2011-11-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Marijuana Abuse
Keywords: cannabis dependence; dronabinol; treatment
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronabinol (Active Comparator): Dronabinol: 20mg bid for a daily maximum dose of 40mg.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if dronabinol decreases the symptoms of marijuana addiction and withdrawal.

DETAILED DESCRIPTION:
Marijuana addiction is associated with significant withdrawal symptoms, including anxiety, irritability, bodily discomfort, and insomnia. The purpose of this study is to determine the effectiveness of dronabinol in reducing withdrawal symptoms.

During this twelve-week, double-blind, placebo-controlled study, study visits will occur twice each week. During study visits, participants will receive either placebo or medication. Throughout the study, all participants will receive individualized psychotherapy sessions. At each study visit, vital signs, self-report ratings, and urine samples will be collected. Participants will have a follow-up evaluation at month 6.

ELIGIBILITY:
Inclusion Criteria:

* men and women between the ages of 18-60
* Meets DSM-IV criteria for current marijuana dependence and reports marijuana as primary drug of abuse
* Individuals must report using marijuana at least 5 days a week and have a marijuana positive urine drug screen on the day of study entry
* Individuals must be capable of giving informed consent and capable of complying with study procedures.
* Women of child-bearing age will be included in the study provided that they are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, blood pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study medication. If a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

* Meets criteria for current psychiatric disorder requiring psychiatric intervention. Disorders that are stable on psychotherapy or pharmacotherapy will not be exclusionary. Individuals will be permitted to take prescribed zolpidem and zaleplon if there is no evidence of dependence on these substances.
* History of seizures
* Known sensitivity to dronabinol
* Unstable medical conditions
* Physical dependence on any other drugs (excluding nicotine) that would require medical detoxification
* Currently taking psychotropic medication with benefit for any other illness than treatment of insomnia
* Pregnant or breast-feeding
* Individuals who have exhibited suicidal or homicidal behavior within the past two years or who have current active suicidal ideation.
* Individuals with coronary vascular disease as indicated by history of abnormal ECG or history of cardiac symptoms.
* Unstable physical disorder which might make participation hazardous such as uncontrolled hypertension (SBP > 150, DBP> 90, or HR > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases < 2-3X upper limit of normal are acceptable), or medically unstable diabetes.
* Subjects in professions in which even mild intoxication would be hazardous (e.g., police officer, bus driver, firefighter).
* Individuals who are court-mandated to treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2005-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

REFERENCES:
- See also: Click here for the Substance Treatment and Abuse Research Service (STARS) website — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were seeking outpatient treatment for problems related to marijuana use and were recruited by local advertising or by clinical referrals in the New York City metropolitan area. Recruitment ran from 3/05-8/09 and patients participated in the trial at a research clinic at Columbia University.
Pre-assignment Details: The trial included a one-week placebo lead-in phase. Individuals who were able to significantly decrease their marijuana use during the first week of the study were not randomized. Participants who reported marijuana use less than twice a week during the placebo lead-in phase were considered placebo responders.
Groups:
- Placebo: Placebo:2 placebo capsules dosed bid for a total of 4 capsules per day
Period: Overall Study
Arm/Group | Dronabinol | Placebo
Started | 79 | 77
Completed | 55 | 44
Not Completed | 24 | 33
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 15 | 19
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 7 | 12
Not completed — non compliant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Placebo | Total
Number analyzed (Participants) | 79 | 77 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (10.8) | 38.4 (9.2) | 37.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 67 | 61 | 128
Region of Enrollment [Number; unit: participants]
  United States | 79 | 77 | 156

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Abstinent From Marijuana During Weeks 7 and 8 of the Trial
Description: Timeline Followback self report data was collected. This daily report was used to assess the proportion of patients abstinent during weeks 7 and 8 of the clinical trial.
Time Frame: weeks 7 and 8
Measure: Number; unit: participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 79 | 77
participants | 14 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were assessed 2x/week for 12 weeks.
Arm/Group | Dronabinol | Placebo
Serious Adverse Events (participants affected / at risk) | 3/79 | 1/77
Other Adverse Events (participants affected / at risk) | 8/79 | 10/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=79) | Placebo (N=77)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — One patient had worsening of chronic asthma that was previously well-controlled, resulting in a brief hospitalization.
diabetes (Endocrine disorders) | 1 (1) | 0 (0) — One patient required hospitalization for worsening diabetes after study completion during the follow-up period.
concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — One patient was involved in an altercation with the police resulting in a hospitalization with eventual discharge.
stomach flu (Gastrointestinal disorders) | 1 (1) | 0 (0) — The fourth patient had a stomach virus and was hospitalized for dehydration and was released after several days.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=79) | Placebo (N=77)
nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 6 (6)
GI upset (Gastrointestinal disorders) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
Consequences of use are often long-term and more subtle. Thus, trying to initiate change over a relatively short period (i.e. patients in the present trial were maintained on the maximum dronabinol dose for only 6 weeks), may have been inadequate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No